CLINICAL TRIAL: NCT02303457
Title: Multicenter, Prospective, Randomized and Controlled Clinical Study 0f CO2 Laser and Open Surgery for T1N0 Glottic Squamous Cell Carcinoma With Anterior Commissure Involved
Brief Title: CO2 Laser and Open Surgery for T1N0 Glottic SCC With Anterior Commissure Involved
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuekui Liu (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Xuekui Liu, chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2014012
Record Dates: First submitted 2014-11-02; First posted 2014-12-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Squamous Cell Carcinoma of Glottis
Keywords: CO2 laser surgery; open surgery; multicenter prospective; randomized; controlled clinical studies; T1N0 squamous cell carcinoma of glottis with anterior commissure involved
MeSH Terms: interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO2 laser surgery (Experimental): CO2 Laser surgery for T1N0 Glottic Squamous Cell Carcinoma With Anterior Commissure Involved. All patients, under general anesthesia, underwent endoscopic excision of the lesion using a carbon dioxide (CO2) laser (Sharplan 100) coupled with a microscope (Zeiss) set to an output power of between 5 and 12 W in superpulse mode. The lesion's resection was accomplished in a radical fashion, with a free margin of 2 mm. For lesions which involved the anterior commissure, the excision plane always uncovered the cartilage.
  Interventions: Procedure: CO2 Laser surgery
- Open surgery (Other): Open Surgery for T1N0 Glottic Squamous Cell Carcinoma With Anterior Commissure Involved.
  open surgery :Frontolateral Vertical Partial Laryngectomy or laryngofissure with cordectomy was accomplished in a radical fashion, with a free margin of 2 mm.
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: CO2 Laser surgery — Patients were randomly assigned to CO2 laser surgery group and open Surgery group.
  Arms: CO2 laser surgery
Procedure: Open Surgery — Patients were randomly assigned to CO2 laser surgery group and open Surgery group.
  Arms: Open surgery

SUMMARY:
Open surgery and CO2 laser surgery are both established treatment modalities for T1N0 glottic carcinoma. It is controversial for T1N0 glottic carcinoma with anterior commissure involved.

ELIGIBILITY:
Inclusion Criteria:

* T1N0 SCC of glottic carcinoma with anterior commissure involve
* No nodal metastasis and distant metastasis
* All patients must have CT/MR and electronic laryngoscope test before surgery and after surgery
* Expected lifetime>1 year
* Patients and families agreed to participate in the test and sign the informed consent
* Without cognitive impairment.

Exclusion Criteria:

* With severe cardiac insufficiency Liver and kidney function is not complete systemic infection patients
* Patients with pregnancy and lactation
* Have surgery contraindications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2014-07; Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
recurrence rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: ye cao, doctor, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China